CLINICAL TRIAL: NCT00345241
Title: Effects of Systane Versus Saline in Maintaining Tear Film Stability at Determined Time Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Vinod Mootha, MD, UTSW Medical Center at Dallas
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 012006-021
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2008-06-23 (Estimated); Status verified 2008-06

CONDITIONS: Keratoconjunctivitis Sicca
Keywords: Blepharitis
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Blepharitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Systane Ocular Drops (OTC)
Drug: Placebo - Saline Drops

SUMMARY:
To evaluate tear film stability of a market lubricant therapeutic eye drop versus saline when using Evaporometry and Interferometry in patients with a diagnosis of Keratoconjunctivitis Sicca (KCS). The purpose of this research is to evaluate evaporative parameters and tear film quality when using Systane lubricating eye drops versus saline in the eyes of dry eye patients at pre-instillation and at 30 and 60 minutes post instillation of drop(s).

DETAILED DESCRIPTION:
The goal of this research is to evaluate and compare the effectiveness of Systane® versus saline on aqueous tear film stability in patients with a diagnosis of Dry Eye Syndrome and to determine the possible application for this product in the future. Systane® is marketed as over-the-counter tear lubricating therapy in the United States under the FDA monograph.

Twelve (12) patients will be enrolled in this two-period crossover, randomized study design. During the course of the study, each patient will be treated with each test articles in the clinic at separate visits. Following the informed consent procedure, a general ocular evaluation, including corneal and conjunctival staining, Schirmer testing, evaporometry, and interferometry assessments will be completed to determine baseline tear evaporation rate. This will occur before any test article is administered to the patient.

Qualified patients will be randomized into two treatment groups. After 1 hour, in order to eliminate any residual sodium fluorescein, patients will be administered one drop of Systane® (40 µl) or saline (40 µl) in each eye per randomization assignment. At 30 and 60 minutes following instillation of drop, evaporometry and interferometry measurements will be repeated again. These tests (pre and post instillation of drops) will be performed in order to establish a comparison for later analysis. The estimated time in completing these visits will be 180 minutes per visit. Patients will be asked to return to the clinic after 2 - 14 days for evaluation of the 2nd assigned treatment.

During the interim study periods, patients will be asked to continue their pre-study routine; using their pre-study ocular lubricant or other tear products at the same frequency. Any changes in the frequency of product use during the interim period or any changes in other concomitant medications will be carefully recorded. This is especially important since many prescription products (e.g., Claritan) have significant effects on lacrimal gland physiology.

An effort will be made to schedule all study visits at approximately the same time of day in order to reduce diurnal variability. For the similar reasons, all patients will be asked not to use any lubricants or ocular medications within one hour of their office visits.

ELIGIBILITY:
Inclusion Criteria: Individuals in good health with signs of Keratoconjunctivitis Sicca are the primary subject population. An ophthalmologist will perform a thorough ocular exam in order to assess entrance qualification into the clinical trial. Patients with apparent Aqueous Tear Deficiency (ATD) with or without slit lamp findings of Meibomian lipid turbidity or difficulty in expression of Meibomian Gland Secretion (MGD) with ocular surface vital staining consistent with ATD in the absence of concurrent disease including lid or ocular surface inflammation beyond 1+ bulbar conjunctival injection will be enrolled.

-

Exclusion Criteria: Patients with active systemic disease or those taking systemic medication that are known to influence AT production will not be considered for this trial. In addition, patients using topical medication who are unable to discontinue them for at least 24 hours prior to baseline evaluation will be excluded as well.

-

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-01; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Evaporametry changes pre and post instillation of test articles in patients with KCS | In Clinic Visit

CONTACTS AND LOCATIONS:
Overall Officials: Harrison D. Cavanagh, M.D., Principal Investigator — University of Texas, Southwestern Medical Center at Dallas
Locations (1):
- University of Texas Southwestern Medical Center at Dallas, Dallas, Texas, United States